CLINICAL TRIAL: NCT02462733
Title: Investigation of the Efficacy of Tools of the Mind for Enhancing Self-Control in Canadian Preschoolers
Brief Title: Efficacy of Tools of the Mind for Enhancing Self-Control in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rosemary Tannock, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000029127
Record Dates: First submitted 2015-05-25; First posted 2015-06-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Self Control; Early Childhood Development
Keywords: Self-control; Preschoolers; Tools of the Mind; Playing to Learn
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tools of the Mind (TOM) (Active Comparator): These 10 classrooms will be exposed to the TOM program.
  Interventions: Behavioral: Tools of the Mind (TOM)
- Playing to Learn (PTL) (Active Comparator): These 10 classrooms will be exposed to the PTL program.
  Interventions: Behavioral: Playing to Learn (PTL)

INTERVENTIONS:
Behavioral: Tools of the Mind (TOM) — TOM is play-based but features explicit, scripted, teacher-directed activities aimed specifically at helping to improve children's self-control skills. Early evidence supports the program efficacy and suggests benefits for children's development more generally (including language, reading and mathematics).
  Arms: Tools of the Mind (TOM)
Behavioral: Playing to Learn (PTL) — PTl is a play based preschool program now in wide use in YMCA childcare settings across Canada (and some in the United States). The activities in PTL are child initiated and are not prescribed. Teachers are trained to observe children at play and to capitalize on learning opportunities as they arise.
  Arms: Playing to Learn (PTL)

SUMMARY:
Self-control has become a strong predictor of academic success and life outcomes. Early childhood development research indicates that greater self-control can lead to better health, greater wealth, and less propensity to engage in criminal activity. This study seeks to assess the strength of the play-based "Tools of the Mind" (TOM) program in improving preschoolers self-control. It will compare TOM to an alternative play-based program, called "Playing to Learn" (PTL), implemented in most YMCA Canada childcare settings across the country. This study hypothesizes that measures of self-control and other measures of social behavior and academic success in preschoolers after two years in the TOM program will be greater than measures of self-control and other measures of social behavior and academic success in preschoolers in the PTL program after two-years.

DETAILED DESCRIPTION:
We will compare growth in self-control and in related areas of development (mathematics, reading, language, social reasoning) in children taught with TOM to children instructed with Playing to Learn (PTL; Eden & Huggins, 2001) - a play based preschool program now in wide use in YMCA childcare settings across Canada (and some in the United States). PTL was developed by an educator/author and by the General Manager of Education, Development, and Research at YMCA Canada. It was selected as the comparison program because it is also a coherent play-based program. In previous studies involving TOM, the comparison programs have differed from TOM on a number of dimensions and often have not been play-based (e.g. Diamond et al., 2007), posing challenges for the interpretation of the results.

In contrast to TOM, the activities in PTL are child initiated and are not prescribed. Teachers are trained to observe children at play and to capitalize on learning opportunities as they arise. For example, children who are using blocks to build a fort, may be encouraged to think about how the size and arrangement of the blocks influences its final structure, to count the number of blocks involved, the number of children the structure can accommodate as well as the structure's affordances. Instruction in self-control is an emergent property of these child-initiated activities. For example, teachers may help children to solve the problem of too few blocks for all of the children interested in the block building activity, by organizing themselves into teams and taking turns. They may assist in conflict resolution by helping children to generate alternative solutions such as stopping to think about the conflict and using words instead of impulsive actions to express their dissatisfaction. Comparison of the development of self-control in children taught with the TOM and PTL programs will thus provide a sense of the benefits (if any) to children of a more focused, teacher-directed approach to teaching self-control.

The primary research question is: Do preschool children taught with the TOM program show greater growth in self-control than their peers who are taught with the PTL program over a two year period? The secondary research question is: If there is a significant difference between the TOM and PTL children in growth in self-control, does that enhanced growth confer benefits for development more generally (for children's cognitive, social, linguistic and academic development)? The proposed efficacy study will be conducted in partnership with the YMCA organization of the greater Toronto area. The study duration will be two years as the TOM program follows a 2-year in-service training plan and children are not expected to reach maximal benefits from exposure to the program until the second year. Twenty YMCA sites will participate, with one participating preschool class (2 teachers) at each site. The criteria for inclusion on the list is that the site must have at least one preschool class, instruction must take place in English, and the preschoolers currently in attendance must not be slated to attend full-day Kindergarten (as per the province's roll out plan) within the study period. Ten sites (classes) will be randomly assigned to either the TOM or the PTL conditions. The YMCA has agreed to provide data on the proportion of families served at each site who pay full fees and those whose fees are subsidized. These data will serve as a proxy for the socioeconomic status of the two groups. Random assignment should result in no difference between the two groups in the mean proportion of families paying full fees.

Both groups of teachers will receive training (TOM) or in-service workshops (PTL) in their respective programs, in each of the two years of the study. Training for TOM will be conducted as required by the program developers; two days of training in the fall and three full days of following up training - one in each in the late fall, winter and spring - of the two years of the study. Professionals from the TOM organization will conduct the TOM training as well as follow-up coaching and assistance to the TOM teachers as needed. Teachers new to the YMCA receive two full days of PTL training. All receive in service workshops every year as well as ongoing in- class teacher training and coaching. The workshops and ongoing assistance are administered by senior YMCA training staff, with a wealth of experience with the PTL program. Every effort will be made to align the amount and the timing of the training/workshops in the two groups. The teachers in both groups will instruct their students according to their assigned programs for the entire study period (2 years), including the summertime.

Program fidelity will be assessed in two ways: 1). using the teacher assessment data generated by experienced evaluators from each program, as per standard practice for both the TOM and PTL programs and 2). by our own classroom observations. Both programs have established methods of assessing teacher fidelity (Bodrova & Leong, 2007; Eden & Huggins, 2001). Successful implementation of the TOM program takes several months to achieve and is said to reach acceptable fidelity levels around March of the first year. Fidelity is assessed periodically, over the first two years of implementation. The YMCA conducts teacher assessments that include PTL fidelity measures annually, around April. We will use the results from the early spring (April) assessments in the two years of the study, for both programs, to determine the teachers' implementation fidelity to their respective programs.

Although both organizations report that reaching acceptable levels of fidelity is not typically problematic, the PTL and TOM assessments will be conducted using different methods, criteria and instruments for documentation. These will capture fidelity to the respective programs - as judged by trained observers from each program - however, they will not address either the differences or possible similarities between programs. This information that could provide critical insights into the mechanisms that might sub-serve different success rates (effects on the development of self-regulation) in the two programs, should such differences arise. Hence, we will also conduct our own observations. A member of our research team will visit each site for a full day and document their observations using a Preschool Observation Measure (POM), which is currently being developed by our research team. The POM contains a list of observable activities and practices one would expect to see in a typical TOM classroom, in a typical PTL classroom and more general practices one would expect to see in any quality child care setting. The observers will rate each classroom with respect to how well the teachers administer these activities. The idea is that TOM teachers should rate more highly on the TOM practices and PTL teachers more highly on the PTL activities, while the two groups may overlap substantially on the more general teaching practices. The observations and ratings will be done in the spring (April - May) of each of the two years of the study.

Participants. Preschool classes and their teachers will be randomly selected from the preschool classrooms at the target sites (n = 10 TOM and 10 PTL classes, 20 TOM and 20 PTL teachers, N= 20 classes and 40 teachers). The criteria for participation in the study for the teachers are: valid Ontario Early Childhood Education certification; permanent, full-time status; no plan to take a leave of absence during the study period; proficiency in spoken English; no known uncorrected hearing or vision impairments; no previous experience with the TOM program; and a signed teacher consent form. As the teachers already provide instruction in English, the English proficiency and no uncorrected impairments requirements are not expected to rule out any teachers currently working at the YMCA.

Twelve to fourteen children, per participating preschool class, will be randomly selected for tracking over the course of the study (n's = 120-140 children in each condition, N = 240-280). Boys and girls will be equally represented. The criteria for student participation are: born between July 2007 and December 2008, inclusive (3 to 4 years of age in 2011), sufficient command of English to understand the teacher's instructions (as judged by their teacher, English as a Second Language - ELL - students will be included provided they meet this criterion); no known uncorrected sensory, neurological, or physical impairments that might prevent full participation in the activities outlined by either program (again, as judged by the teacher) and a signed parental consent form. We will obtain information regarding the above teacher and student criteria from the YMCA.

As our primary research question concerns the relative efficacy of TOM for improving self-regulation skills, the primary outcome measures will be two tasks that tap inhibitory control (see below). Our secondary research question concerns the implications for enhancing self-control for children's development more generally including their cognitive, social/emotional, language, and academic development as well their attention skills and overall adjustment. Accordingly, we will measure change over the study period in the development of children's classroom and home behaviour, attention skills, theory of mind, receptive and expressive vocabulary, mathematics, as well as drawing, writing and pre/early literacy skills, all of which have been linked to executive function (see e.g. McInnes, Humphries, Hogg-Johnson & Tannock, 2003 and Martinussen, Hayden, Hogg-Johnson & Tannock, 2005, for poor attention skills and Attention Deficit Hyperactivity Disorder (ADHD); Kyte, Goodyer & Sahakian, 2005 for inhibitory control and depression; Carlson & Moses, 2001 for theory of mind and executive function; Carlson & Moses, 2001 and Hughes, 1998 for inhibitory control and language, and Blair & Razza, 2007 and Bull & Scerif, 2001 for inhibitory control and reading and mathematics skills). All of the measures will be administered in the fall and the spring of the two years of the study (2011-2012 and 2012-2013).

Children will be tested individually, in a quiet location in their preschool, during regular preschool hours. We will coordinate with the teachers to ensure minimal disruption to their classrooms during the four data collection time points. The total test time for the children is 35-45 minutes at each time point (spring and fall of the two study years), which will be divided into two test sessions of about 25 minutes each (excluding the time for the drawings/play plans which will be administered as part of the PTL and TOM curricula). To help maintain motivation, the tasks will be presented in the form of games, breaks will be given between tasks as needed and children will be praised for their efforts. Previous experience has shown that children in this age group find such "games" highly enjoyable and that 30 minutes of focused attention to a variety of tasks is well within the attention range of most preschoolers, when working with experienced experimenters.

ELIGIBILITY:
Inclusion Criteria:

* Born between July 2007 and December 2008, inclusive (3 to 4 years of age in 2011)
* Sufficient command of English to understand the teacher's instructions (as judged by their teacher, English as a Second Language - ELL - students will be included provided they meet this criterion)
* Signed parental consent form

Exclusion Criteria:

* Known uncorrected sensory, neurological, or physical impairments that might prevent full participation in the activities outlined by either program (again, as judged by the teacher)
* Insufficient command of English
* No parental consent given

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Inhibitory Control | Change from baseline to 18 months
  Inhibitory Control will be measured through the Day/Night task (Gerstadt et al., 1994). Children are presented with a white card depicting a yellow sun and a black card depicting a white moon and stars. They are then instructed to play a "silly" game in which they must say "day" when they see the night card and "night" when they see the day card. Hence, they must inhibit the pre potent response to say the word that is associated with the picture, and say the opposite word. Children receive 16 test trials in which the cards are presented in a fixed pseudorandom order. There are no breaks or rule reminders. Day/Night is a well-established and widely used task, ubiquitous in the developmental and developmental neuroscience literature. The task takes less than 5 minutes to complete.task.

SECONDARY OUTCOMES:
Early Childhood Development - Theory of Mind | Change from baseline to 18 months
  Children will receive a version of the standard false belief task (Wimmer & Perner, 1983). False belief tasks tap inhibitory control and perspective taking in a social context, fundamental skills for establishing successful relationships.
Early Childhood Development - Language | Change from baseline to 18 months
  Children's receptive and expressive vocabulary will be measured with the Peabody Picture Vocabulary Test (PPVT-R; Dunn & Dunn, 1981) and the Expressive One Word Picture Vocabulary Test (EOWPVT - R; Brownell, 2000), respectively. For the PPVT, children are presented with a matrix of four pictures on each trial and required to point to the picture that goes with a word the experimenter says aloud.
Early Childhood Development - Reading | Change from baseline to 18 months
  Pre/early reading skills will be assessed with Get Ready to Read (GRTR; Whitehurst & Lonigan, 2001) a screening tool designed to assess progress in developing early literacy skills in preschoolers.
Early Childhood Development - Mathematics | Change from baseline to 18 months
  Children's emerging number sense will be assessed with the "Point to X" task (PTX; Wynn, 1992). PTX assesses children's conceptual understanding of counting, as opposed to their rote knowledge of counting terms. Children will be required to point to the correct one of two arrays, each depicting a different number of squares, that shows the number of squares corresponding to a number the experimenter says aloud.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ferguson, MD, Principal Investigator — The Hospital for Sick Children; Tracy Solomon, MD, Principal Investigator — The Hospital for Sick Children; Rosemary Tannock, MD, Principal Investigator — OISE, University of Toronto
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No